CLINICAL TRIAL: NCT00944879
Title: Preparing for Adolescent HIV Vaccine Trials in South Africa: a Multi-centre Study to Evaluate Acceptability of the HPV Vaccine in Adolescents
Brief Title: Preparing for Adolescent HIV Vaccine Trials in South Africa:
Acronym: CATSA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Desmond Tutu HIV Centre (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Professor Linda-Gail Bekker, Desmond Tutu HIV Centre
Other Study IDs: 35384; CT.2006.33111.004
Record Dates: First submitted 2009-07-20; First posted 2009-07-23 (Estimated); Last update posted 2009-08-17 (Estimated); Status verified 2009-07

CONDITIONS: HIV Infection; HIV Infections
Keywords: HIV; vaccine; prevention; HPV; adolescents
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood for HIV, syphilis and pregnancy testing
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- HPV vaccine: Those choosing to receive the HPV vaccine
- no HPV vaccine: Those choosing not to receive the HPV vaccine

SUMMARY:
This study will use the licensed HPV vaccine, Gardasil, as a surrogate for an HIV vaccine, in order to explore some of the ethico-legal,psycho-social and logistical challenges involved in running an HIV vaccine trial in adolescents.

DETAILED DESCRIPTION:
This study will use the licensed HPV vaccine, an alternative STI vaccine, as a proxy for an HIV vaccine and thereby identify potential challenges to the inclusion of adolescents in HIV prevention trials. The study will allow for site capacity building in terms of recruiting and retaining an HIV-negative high-risk adolescent cohort, and assessing the acceptability of an STI vaccine to adolescents and their parents or guardians. Correlates of vaccine uptake, refusal, retention and attrition will be determined. In addition, the study will document the incidence of HIV, other sexually transmitted infections (STI's) and pregnancies and circumcisions in this age group. Different methods of assessing understanding in adolescents will be tested, to ensure that informed consent is being achieved. Experiences of privacy and confidentiality issues for adolescents in such research will be explored. Finally, psycho-social correlates of sexual risk and protective behaviour will be examined.

The study is designed as a longitudinal cohort study with a self-selected intervention and control group. Adolescents and parents will be recruited through community outreach and invited to attend a Vaccine Discussion Group (VDG) to learn more about the HPV vaccine. Parental/ legal guardian consent and adolescent assent will be obtained prior to screening. After screening to ensure volunteers meet inclusion criteria, 1400 participants will be enrolled across seven sites. At this point, they will decide whether or not they want to receive the HPV vaccine. Those who do will receive three doses, at 0, 2 and 6 months. All participants will undergo HIV and pregnancy testing, receive risk reduction counseling and complete questionnaires at 0, 2, 6 and 9 months. Recruitment and retention will be monitored and data as described above will be collected throughout the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Youth age 12-17 years
* For 12-15 year olds - no sexual risk criteria
* For 16-17 year olds (the age of lawful consent to sex in South Africa): sexually active (ever had sexual intercourse)
* Willing to participate in HIV testing and counseling
* Willing and able to assent to study
* Parent or legal guardian willing to provide written consent
* HIV-negative serostatus at screening and enrolment
* Females must have a negative pregnancy test at screening/enrolment
* Females must not be breastfeeding

  * Additional inclusion criteria for those accepting HPV vaccination:
* No HPV immunizations
* Females should agree to avoid pregnancy through to the end of the study and to take contraceptives throughout the study (access provided)

Exclusion Criteria:

* Exclusion criteria for those accepting HPV vaccination:

  * Presence of any serious illness requiring treatment with systemic medications, excluding short course oral steroids or inhaled steroid treatment for asthma
  * Contra-indication to vaccination, such as bleeding disorder
  * Previous allergic reaction to any vaccines or to constituents of these vaccines (yeast, thimerosal or aluminum)
  * Current immunomodulator therapy
  * Receipt of immunosuppressor therapy (more than 10mg/day of prednisone or equivalent for >1 week) in the 6 months preceding enrollment date
  * Receipt of any vaccine within two weeks preceding enrollment date

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: South African adolescents aged 12 to 17
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Recruitment and retention | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Linda-Gail Bekker, MBChB PhD, Principal Investigator — Desmond Tutu HIV Centre
Locations (1):
- Desmond Tutu HIV Centre, Cape Town, South Africa